CLINICAL TRIAL: NCT03853200
Title: In-vivo Comparison of Antibacterial Efficacy of Three Different Solutions as Final Irrigant During Endodontic Therapy: A Randomized Controlled Trial
Brief Title: Comparison of Antibacterial Efficacy of Three Final Irrigants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Hasan Afaq Zaidi, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-796/DUHS/Approval/2016/324
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Endodontic Disease; Root Canal Infection
Keywords: Final irrigation; Irrigation in Endodontics; QMix; CFU; Colony forming unit; MRS; Microbiological root canal sampling
MeSH Terms: conditions — Dental Pulp Diseases | interventions — QMix root canal irrigant; Edetic Acid; Chlorhexidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group I (Experimental): QMix the solution under investigation which includes CHX EDTA and detergent QMix Root Canal Irrigant
  Interventions: Drug: QMix Root Canal Irrigant
- Group II (Active Comparator): it involves use of two irrigant solutions, 17%EDTA+2%Chlorhexidine
  Interventions: Drug: 17%EDTA+2%Chlorhexidine
- Group III (Active Comparator): 17% EDTA with no antibacterial activity . the control group
  Interventions: Other: EDTA

INTERVENTIONS:
Drug: QMix Root Canal Irrigant — Endodontic irrigant recommended for final irrigation
  Other Names: QMIx
  Arms: Group I
Drug: 17%EDTA+2%Chlorhexidine — two endodontic irrigants will be used in this group in a sequential manner
  Other Names: EDTA; Chlorhexidine
  Arms: Group II
Other: EDTA — 17% EDTA irrigation solution
  Other Names: Ethylenediaminetetra acetic acid
  Arms: Group III

SUMMARY:
This study was conducted to determine the antibacterial affect of three different solutions used as final irrigant during endodontic therapy. The investigator's objective was to compare the antibacterial affect of relatively new final irrigant QMix with EDTA and Qmix with EDTA+CHX by evaluating the bacteriological status of the root canal before and after use of the final irrigant.

DETAILED DESCRIPTION:
The aim of this clinical trial is to compare the antibacterial efficacy of Qmix, to 17% EDTA+ Chlorhexidine and 17% EDTA, used as final irrigants, during endodontic procedure.

Endodontic treatment was carried out on 90 necrosed teeth of patients under rubber dam isolation and strict sterilization protocol. The teeth were divided into three groups; A, B and C depending on the type of final irrigant to be used. The chemo-mechanical preparation of all the 90 samples was carried out using ProTaper Universal (Dentsply) File system, and 3% sodium Hypochlorite. All the samples from each group were then irrigated according to the final rinse protocol (FRP). Group A was irrigated with Qmix; Group B with 17% EDTA + 2% Chlorhexidine and Group C (Control group) 17% EDTA.

Three bacteriologic samples were taken during the procedure from each root canal under study in all three groups, using sterile paper points. Sample A was collected after access cavity opening and negotiation of the canal but before chemo-mechanical preparation. Sample B was taken after chemo-mechanical preparation but before the use of the final irrigant. Sample C was collected after the use of final irrigation solution. The samples were collected with sterile paper points and were then transferred to microbiology laboratory in microtubes containing Brain Heart Infusion (BHI) broth within 2 hours of sample collection for obtaining the colony forming unit (CFU) counts.

ELIGIBILITY:
Inclusion Criteria:

* Teeth:

  * Single rooted (One root canal)
  * Necrosed teeth requiring root canal treatment.
  * Teeth with mature apices
  * Permanent dentition
  * Mandibular & Maxillary
  * PAI category 1 to 4

Exclusion Criteria:

• Teeth:

* Single rooted teeth with multiple canals
* Root canal treated
* Requiring elective endodontic therapy
* With partial necrosis
* Fractured
* Having calcified and obliterated canals.
* Having root resorption
* Root canals which could not be negotiated to full working length with #10 K file
* Having severe periodontitis with exacerbating features (PAI = 5)
* Having grade III mobility
* Patients who took systemic antibiotics in past four weeks.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Colony forming Unit | Before and after use of final irrigant, up to 5 minutes
  Change in the Colony forming unit (CFU) of the root canal sample will be assessed by determining the difference between Mean CFU of sample taken before use of final irrigant and sample taken after use of final irrigant.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Zaidi, BDS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Hasan Zaidi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided